CLINICAL TRIAL: NCT04229433
Title: A Phase I, Randomized, Single -Blind, Placebo-Controlled, Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR2285 Tablets in Healthy Subjects
Brief Title: The Multiple Dose of PK/PD Study of SHR2285 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHR2285-102
Record Dates: First submitted 2019-12-18; First posted 2020-01-18 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2020-01

CONDITIONS: Thrombus
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Intervention Model Description: Multiple dose of PK/PD Study of SHR2285 Tablets in Healthy Subjects
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR2285 (Experimental): Participants received one of 3 dose levels of SHR2285 administered as multiple oral doses.
  Interventions: Drug: SHR2285 tablet; Drug: Placebo
- Placebo (Experimental): Participants received one of 3 dose levels of placebo administered as multiple oral doses.
  Interventions: Drug: SHR2285 tablet; Drug: Placebo

INTERVENTIONS:
Drug: SHR2285 tablet — Pharmaceutical form: SHR2285 tablet Route of administration: single dose and multiple doses.
Drug: Placebo — Pharmaceutical form: Placebo tablet Route of administration: single dose and multiple doses.

SUMMARY:
The study is a randomized, single-blind, placebo-controlled, multiple-dose escalation Phase I trials. 2 dose groups were designed, 12 subjects in each dose group.The drug was administered single dose and multiple doses.

ELIGIBILITY:
Inclusion Criteria:

1. males or females, aged 18-45.
2. subjects with no cardiovascular disease, sitting blood pressure: 90mmHg ≤SBP<140mmHg; 50mmHg ≤DBP<90mmHg and 50 ≤ HR <110 beats / min.
3. body mass index (BMI) between 18 to 28.
4. Participant in general good health. No clinically significant findings in vital signs, physical examination, 12-lead ECG ,X-ray and laboratory parameters.

Exclusion Criteria:

1. males or females, aged 18-45.
2. subjects with no cardiovascular disease, sitting blood pressure: 90mmHg ≤SBP<140mmHg; 50mmHg ≤DBP<90mmHg and 50 ≤ HR <110 beats / min.
3. body mass index (BMI) between 18 to 28.
4. Participant in general good health. No clinically significant findings in vital signs, physical examination, 12-lead ECG ,X-ray and laboratory parameters.

Exclusion Criteria:

1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin/direct bilirubin > 1X ULN during screening/baseline.
2. Serum creatinine> 1X ULN during screening/baseline.
3. Abnormal coagulation function.
4. A clinical history of coagulation dysfunction; subjects with adverse reaction of antiplatelet drugs or anticoagulant drugs.
5. Subjects with severe head trauma or head surgery within 2 years or surgery within 3 months prior to the screening.
6. Blood donation or blood loss within 1 month≥200 mLor≥400 mL within 3 months before administration.
7. Human immunodeficiency virus antibody (HIV-ab), syphilis serological examination, hepatitis b virus surface antigen (HBsAg), hepatitis c virus antibody (HCV-ab) were positive.

8.3 months prior to screening involved in any drug or medical device clinical studies or within 5 half-life of drugs before screening.

9.Female subjects who did not receive contraception at least 30 days before administration.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2020-11-08 (Actual); Study Completion 2020-11-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events and serious adverse events. | Pre-dose to 7 days after multiple dose administration.

SECONDARY OUTCOMES:
PK parameter will be evaluated. | Pre-dose to 3 days after single dose administration
  Area under the plasma concentration versus time curve (AUC) for single dose of SHR2285.
Maximum observed serum concentration (Cmax) for single dose of SHR2285. | Pre-dose to 3 days after single dose administration
Time to maximum observed serum concentration (Tmax) for single dose of SHR2285. | Pre-dose to 3 days after single dose administration
Apparent total clearance of the drug from plasma after oral administration (CL/F) for single dose of SHR2285. | Pre-dose to 3 days after single dose administration.
Apparent volume of distribution after non-intravenous administration (V/F) for single dose of SHR2285 | Pre-dose to 3 days after single dose administration.
Time to elimination half-life (T1/2) for single dose of SHR2285. | Pre-dose to 3 days after single dose administration
Area under the plasma concentration versus time curve (AUC) for multiple dose of SHR2285. | Pre-dose to 2 days after multiple dose administration
Steady-state peak concentration (Cmax，ss) for multiple dose of SHR2285. | Pre-dose to 2 days after multiple dose administration
Steady state valley concentration (Ctrough，ss) for multiple dose of SHR2285. | Pre-dose to 2 days after multiple dose administration
Time to maximum observed serum concentration (Tmax) for multiple dose of SHR2285. | Pre-dose to 2 days after multiple dose administration.
Time to elimination half-life (T1/2) for multiple dose of SHR2285. | Pre-dose to 2 days after multiple dose administration
Steady-state apparent total clearance of the drug from plasma after oral administration (CLSS/F) for multiple dose of SHR2285. | Pre-dose to 2 days after multiple dose administration.
Steady-state apparent volume of distribution after non-intravenous administration (VSS/F) for multiple dose of SHR2285. | Pre-dose to 2 days after multiple dose administration.
Accumulation ratio (Racc) for multiple dose of SHR2285. | Pre-dose to 2 days after multiple dose administration.
Percentage of fluctuation (PTF%) for multiple dose of SHR2285. | Pre-dose to 2 days after multiple dose administration.
PD parameter will be evaluated. | Pre-dose to 3 days after single dose administration.
  FXI activity; Change of APTT, PT, INR from baseline.
PD parameter will be evaluated. | Pre-dose to 2 days after multiple dose administration.
  FXI activity; Change of APTT, PT, INR from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejing Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided